CLINICAL TRIAL: NCT07174167
Title: Effectiveness of Genicular Nerve Block on Pain and Disability in Chronic Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Genicular Nerve Block in Chronic Knee Osteoarthritis
Acronym: GNB-KOA-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Gunay, MD, Medical Doctor, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK 2023/58
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Gonarthrosis; Primary; Genicular Nerve Block; Gonarthritis
Keywords: genicular nerve block; knee osteoarthritis; pain; disability; gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Prilocaine; Triamcinolone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- genicular nerve block with local anesthetic (Active Comparator): Group 1 (GNB with local anesthetic only): Patients received a genicular nerve block (GNB) with 6 mL of 2% prilocaine and participated in a knee exercise program.
  Interventions: Drug: Genicular nerve block with prilocaine
- genicular nerve block with local anesthetic and corticosteroid (Active Comparator): Group 2 (GNB with local anesthetic and corticosteroid): Patients received GNB with 5 mL of 2% prilocaine in combination with 1 mL/40 mg of triamcinolone and followed the same exercise regimen.
  Interventions: Drug: genicular nerve block with prilocaine and triamcinolone
- sham injection with saline (Sham Comparator): Group 3 (Control group): Patients received a placebo injection (6 mL of 0.9% saline) with the knee exercise program.
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Genicular nerve block with prilocaine — ultrasound guided genicular nerve block (GNB) injecting 6 mL of 2% prilocaine to the genicular nerves
  Other Names: group 1
  Arms: genicular nerve block with local anesthetic
Drug: genicular nerve block with prilocaine and triamcinolone — ultrasound guided genicular nerve block (GNB) injecting 5 mL of 2% prilocaine in combination with 1 mL/40 mg of triamcinolone to the genicular nerves
  Other Names: group 2
  Arms: genicular nerve block with local anesthetic and corticosteroid
Drug: Sham injection — placebo injection using 6 mL of 0.9% saline to knee region other than genicular nerves
  Other Names: group 3
  Arms: sham injection with saline

SUMMARY:
The goal of this clinical trial is to evaluate whether genicular nerve block (GNB) is effective in reducing pain in patients with knee osteoarthritis. It will also assess the comparative efficacy of different injection protocols.

The main questions it aims to answer are:

Does genicular nerve block with corticosteroid and local anesthetic provide superior pain relief compared with local anesthetic alone or placebo?

Are there differences in clinical outcomes between the three treatment groups?

Researchers will compare three groups:

GNB with corticosteroid plus local anesthetic

GNB with local anesthetic alone

Sham procedure with saline (placebo control)

Participants will:

Receive the assigned injection protocol in accordance with their group

Be evaluated at baseline and scheduled follow-up visits for pain intensity and functional status

Report their pain scores and functional limitations using standardized assessment tools

ELIGIBILITY:
Inclusion Criteria:

* age between 45 and 75
* diagnosed with knee osteoarthritis (OA) according to the American College of Rheumatology (ACR) criteria
* possessing a Kellgren-Lawrence radiological grade of 2-3

Exclusion Criteria:

* any joint injection to the target knee in the past 3 months
* physical therapy for the target knee within the last 3 months
* previous knee surgery
* inflammatory rheumatic diseases
* active lumbar radiculopathy on the same side
* neurological disorders (e.g., Alzheimer's or dementia)
* uncontrolled cardiopulmonary diseases
* pregnancy or lactation
* obesity (body mass index [BMI] >35)
* presence of a pacemaker
* active malignancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | at baseline, 1 week, and 1 month after treatment
  Visual Analog Scale (VAS): The VAS assesses pain intensity on a 10-centimeter scale. Patients indicate their pain levels using two verbal descriptors at the end of each scale.

SECONDARY OUTCOMES:
Functional status using WOMAC | baseline, 1 week, and 1 month after treatment
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire assessed pain and disability.
Functional status using 40-Meter Fast Walking Test | at baseline, 1 week, and 1 month after treatment
  40-Meter Fast Walking Test: This test involved a designated 10-meter walking track. Patients walked at their maximum pace for four laps. No warm-up was conducted, and the time spent turning at the lines was excluded from the calculation
Pressure Pain Threshold (PPT) | baseline, 1 week, and 1 month after treatment
  Pressure Pain Threshold (PPT): The Commander Algometer (JTECH Medical, Utah, USA) was utilized to measure PPT at both the medial and lateral sides of the patella. The probe tip of the algometer was applied perpendicularly to the skin, and pressure was gradually increased. Patients indicated when they first experienced discomfort, at which point the measurement was recorded. This procedure was repeated three times, and the average value was noted.

OTHER OUTCOMES:
Ultrasound evaluation | baseline
  Ultrasound measurements were taken to assess patellofemoral cartilage thickness and quadriceps muscle thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study data are available with the researcher and can be provided to the relevant authorities if required.

REFERENCES:
- [Background] Li W, Xu F, Chen F, Cao L, Bao X. Effect of Genicular Nerve Block (GNB) on Pain in Lesions of the Knee Joint: A Meta-Analysis of Randomized Controlled Trials. J Pain Res. 2025 Jan 30;18:511-522. doi: 10.2147/JPR.S503937. eCollection 2025. PMID 39901967
- [Background] Kim DH, Lee MS, Lee S, Yoon SH, Shin JW, Choi SS. A Prospective Randomized Comparison of the Efficacy of Ultrasound- vs Fluoroscopy-Guided Genicular Nerve Block for Chronic Knee Osteoarthritis. Pain Physician. 2019 Mar;22(2):139-146. PMID 30921977
- [Background] Kim DH, Choi SS, Yoon SH, Lee SH, Seo DK, Lee IG, Choi WJ, Shin JW. Ultrasound-Guided Genicular Nerve Block for Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial of Local Anesthetic Alone or in Combination with Corticosteroid. Pain Physician. 2018 Jan;21(1):41-52. PMID 29357330
- [Background] Shanahan EM, Robinson L, Lyne S, Woodman R, Cai F, Dissanayake K, Paddick K, Cheung G, Voyvodic F. Genicular Nerve Block for Pain Management in Patients With Knee Osteoarthritis: A Randomized Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):201-209. doi: 10.1002/art.42384. Epub 2022 Nov 11. PMID 36369781